CLINICAL TRIAL: NCT04452708
Title: The Safety of High Flow Nasal Cannula and Noninvasive Ventilation for Treatment of Patients With COVID-19 Complicated by Respiratory Failure
Brief Title: HFNC and NIV for COVID-19 Complicated by Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Other Study IDs: 2020.203
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Failure
Keywords: HFNC; NIV; oxygen; COVID-19
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NIOSH air samplers are located around the sampling bed ('Centre'), on the side of the sampling bed ('Side'), or relocated during the period of the sampling and application of each respiratory therapy. Air is collected at 3.5L/minute into three size fractions: >4μm (collected in a 15ml tube), 1-4μm (1.5ml tube) and <1μm (by a polytetrafluoroethylene (PTFE) membrane filter with 3.0μm pore size). All the tubes are then transported to the laboratory at 4°C, vortexed, and the VTM is aliquoted and stored at -80°C for subsequent laboratory analysis by RT-PCR. Viral loads will be measured from the patient's upper respiratory tract (nasopharyngeal flocked swab and throat swab) on admission and serially second daily during hospitalization by means of quantitative RT-PCR assay.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFNC at 30-60L/min: HFNC at 50-60L/min with humidification at 37C (Airvo 2, Fisher & Paykel, Auckland, New Zealand) will be applied for patients with moderate type 1 respiratory failure
  Interventions: Device: HFNC
- NIV: NIV (Respironics V60) via oronasal mask (Quattro, ResMed) will be reserved for patients with type 2 respiratory failure
- Conventional nasal oxygen: Oxygen 1-5 L/min via nasal cannula for those with mild type 1 respiratory failure

INTERVENTIONS:
Device: HFNC — HFNV vs NIV vs conventional nasal cannula
  Other Names: NIV; Conventional nasal cannula
  Groups: HFNC at 30-60L/min

SUMMARY:
Background: Patients with COVID-19 have a range of clinical spectrum from asymptomatic infection, mild illness, moderate infection requiring supplemental oxygen and severe infection requiring intensive care support. High flow nasal cannula (HFNC) oxygen therapy and noninvasive ventilation (NIV) may offer respiratory support to patients with COVID-19 complicated by acute hypoxemic respiratory failure if conventional oxygen therapy (COT) fails to maintain satisfactory oxygenation but whether these respiratory therapies would lead to airborne viral transmission is unknown.

Aims: This study examines whether SARS-2 virus can be detected in small particles in the hospital isolation rooms in patients who receive a) HFNC, b) NIV via oronasal masks and c) conventional nasal cannula for respiratory failure.

Method: A field test to be performed at the Prince of Wales hospital ward 12C single bed isolation room with 12 air changes/hr on patients (n=5 for each category of respiratory therapy) with confirmed COVID-19 who require treatment for respiratory failure with a) HFNC up to 60L/min, b) NIV via oronasal masks and c) conventional nasal cannula up to 5L/min of oxygen. While the patient is on respiratory support, we would position 3 stationary devices in the isolation room (one next to each side of the bed and another at the end of the bed) of the patient with confirmed COVID-19 infection, and sample the air for four hours continuously.

Results & implications: If air sampling RTPCR and viral culture is positive, this would objectively confirm that HFNC and NIV require airborne precaution by healthcare workers during application.

DETAILED DESCRIPTION:
A novel coronavirus, subsequently named by the World Health Organization (WHO) as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), emerged as the cause of atypical pneumonia linked to a seafood market in Wuhan, China in Dec 2019. Since then, SARS-CoV-2 related-disease (named COVID-19 by the WHO), has spread internationally to the scale of a global pandemic. Although most patients present with mild respiratory symptoms, some have severe pneumonia and a small proportion may become critically ill. Severe COVID-19 disease often progresses to acute hypoxemic respiratory failure requiring high fractional concentration of inspired oxygen (FiO2) and consideration for non-invasive ventilation (NIV) strategies.

High-flow nasal cannula (HFNC) has emerged as a non-invasive strategy improving oxygenation and carbon dioxide clearance by, in comparisons to other NIV strategies, better matching patients' inspiratory demands by delivering up to 60 L/min of gas flow and FiO2 up to 1.0. A systematic review found low certainty evidence suggesting benefit of HFNC in reducing the need for invasive mechanical ventilation (IMV) or escalation of oxygen therapy compared to conventional oxygen therapy (COT), and moderate certainty evidence suggesting no large difference in mortality. HFNC may reduce the need for IMV and associated complications such as ventilator-associated pneumonias, and alleviate the strain on healthcare systems during the COVID-19 pandemic.

COVID-19 spreads predominantly through respiratory droplets and fomites. There is concern, however, that airborne transmission may occur during respiratory procedures that generate aerosols. Airborne transmission involves smaller particles, typically <5μm in diameter, which may remain suspended in the air for extended periods of time, transmitted over distances greater than 1m, and inhaled into the lower airways. Reduction of respiratory particles to <5 µm involves evaporation of larger droplets and their contained organisms, and rehydration after deposition into the airway; therefore, airborne transmission is organism-specific, and requires the organism to survive a process of desiccation and aerosolization in sufficient numbers to cause infection. SARS-CoV2 has been shown to survive in air for 3 hrs after deliberate aerolization.

The Surviving Sepsis Campaign (SSC) COVID-19 guidelines provide a weak recommendation for the preferential use of HFNC over other NIV strategies in patients refractory to COT for type 1 respiratory failure.10 The use of high flow rates raises concerns that HFNC may cause aerosolization of infectious particles. Using a human patient simulator and smoke particles as markers visualized by a laser light sheet, HFNC with humidification may disperse exhaled air up to 172mm upward and 620mm laterally when the nasal cannula is clipped on properly and loosely respectively. Using the same methodology, NIV via the old generation oronasal masks could disperse exhaled air diffusely but there is limited exhaled air dispersion through the new generation masks with better design of the exhalation ports. In contrast, exhaled air dispersion from conventional nasal cannula delivering oxygen at 5L/min without humidification may disperse exhaled air to 1m towards the end of the bed.

Due to lack of field data on the use of these respiratory therapies in patients with COVID-19 complicated by respiratory failure, the role of fine particle aerosols in transmission of viral infection during application of HFNC and NIV is unknown. Because of uncertainty around the potential for aerosolization, the WHO has recommended that HFNC, NIV, including bubble CPAP, should be used with airborne precautions until further evaluation of safety can be completed. To alleviate concern by the healthcare workers in delivering these respiratory therapies to patients with COVID-19 complicated by respiratory failure, it is important to conduct a field test using viral samplers in patients with COVID-19 who require these therapies for respiratory failure.

Aims and objectives This study aims to detect whether SARS-2 virus can be detected in small particles in the hospital isolation rooms in patients who receive a) HFNC up to 60L/min, b) NIV via oronasal masks and c) conventional nasal cannula.

Subjects and indications of respiratory therapy:

This is a field test to be performed at the Prince of Wales hospital ward 12C single bed isolation room with 12 air changes per hr on patients (n=5 for each category of respiratory therapy) with confirmed COVID-19 who require treatment for respiratory failure with a) HFNC up to 60L/min, b) NIV via oronasal masks and c) conventional nasal cannula up to 5L/min of oxygen. Five patients in each treatment category will be recruited as the majority (80%) of confirmed cases in HK have been mild without respiratory failure. For example, among the 974 cases as of 10 April 2020, 23 and 25 patients respectively have ever required supplemental oxygen at least 3L/min on the isolation wards and ICU support (for IMV, ECMO or shock). Different respiratory therapy will be decided by the physician on duty for patients with different degree of respiratory failure. In general, conventional nasal cannula is used for mild respiratory failure while HFNC is required to those who remain hypoxic. NIV is usually applied for those with type 2 respiratory failure. In adults with COVID-19, the SSC Guidelines suggest starting supplemental oxygen if the peripheral oxygen saturation (SPO2) is < 92% (weak recommendation, low quality evidence), and recommend starting supplemental oxygen if SpO2 is < 90% (strong recommendation, moderate quality evidence) to achieve SpO2 not higher than 96%. For adults with COVID-19 and acute hypoxemic respiratory failure despite COT, the SSC guidelines suggest using HFNC over NIV (weak recommendation, low quality evidence). In adults with COVID-19 and acute hypoxemic respiratory failure, if HFNC is not available and there is no urgent indication for endotracheal intubation, the SSC guidelines suggest a trial of NIV with close monitoring and short-interval assessment for worsening of respiratory failure (weak recommendation, very low quality evidence).

Respiratory therapy: COT with nasal cannula 1-5L/min of oxygen will be used to maintain SpO2 around 95% for patients with type 1 respiratory failure. If this is not achievable despite 5L/min of oxygen, HFNC at 50-60L/min with humidification at 37C (Airvo 2, Fisher & Paykel, Auckland, New Zealand) will be applied while NIV (Respironics V60) via oronasal mask (Quattro, ResMed) will be reserved for patients with type 2 respiratory failure.

Air samplings:

On each air sampling period while the patient is on respiratory support, we would position 3 stationary devices in the isolation room (one next to each side of the bed and another at the end of the bed) of the patient with confirmed COVID-19 infection, and sample the air for four hours continuously. The National Institute for Occupational Safety and Health (NIOSH) device consists of a three-stage cyclone air samplers set at height 1.5m and 1.0m, which represent the mouth heights of a standing and sitting adult respectively and a meter that records temperature and relative humidity (at height 1.3m) every four minutes. The NIOSH samplers are located around the sampling bed ('Centre'), on the side of the sampling bed ('Side'), or relocated during the period of the sampling. The NIOSH samplers are placed in the range of 0.5-1m (when placed next to the sampling bed) to 2-2.5m from the patient's head when placed at the end of the bed.

Air is collected at 3.5L/minute into three size fractions: >4μm (collected in a 15ml tube), 1-4μm (1.5ml tube) and <1μm (by a polytetrafluoroethylene (PTFE) membrane filter with 3.0μm pore size). For five sampling runs, an extra air sampler (set at height 0.8m) unconnected to a pump will be added to the device as a negative control. After each collection, the 15ml and 1.5ml tubes are detached and 1 ml of viral transport medium (VTM) are added. The filter is removed and immersed in 1mL of VTM inside a 5ml tube. All the tubes are then transported to the laboratory at 4°C, vortexed, and the VTM is aliquoted and stored at -80°C for subsequent laboratory analysis by reverse-transcriptase-polymerase-chain-reaction (RT-PCR). New sampling tubes and filters are used and the samplers and other equipment are disinfected between uses. The tripod, air tubing, sound-proof box and the meter are disinfected with Med-Clean (M&W International Ltd., Hong Kong), the NIOSH air samplers with 1% Virkon and 2% Citranox (Alconox Inc, NY, USA), and the filter cassettes are autoclaved.

Viral loads:

Viral loads will be measured from the patient's upper respiratory tract (nasopharyngeal flocked swab and throat swab) on admission and serially second daily during hospitalization by means of quantitative RT-PCR assay with primers and probes targeting the N and Orf1b genes of SARS-CoV-2.

Data processing and analysis:

Statistical analysis: Dependent variables are identified as the nasopharyngeal flocked swab and throat swab viral load (log10 copies/mL) and detection of viral RNA from one or more participant air samples (positive) vs. all negative air samples. The Wilcoxon-Mann-Whitney, Kruskal Wallis tests and Spearman correlation are used to assess the presence of statistically significant correlations or distributions between independent variables and the upper respiratory tract swab viral load, while the Wilcoxon-Mann-Whitney and Fisher's exact tests are used for air samples. Statistical analysis was performed using SAS University Edition (SAS Institute, Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria: Patients with confirmed COVID-19 who require treatment for respiratory failure

Exclusion Criteria:

* inability to provide consent;
* severe respiratory failure requiring invasive ventilatory support;
* septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a field test being conducted at the Prince of Wales hospital ward 12C single bed isolation room with 12 air changes per hr on patients (n=5 for each category of respiratory therapy) with confirmed COVID-19 who require treatment for respiratory failure with a) HFNC up to 60L/min, b) NIV via oronasal masks and c) conventional nasal cannula up to 5L/min of oxygen. Five patients in each treatment category will be recruited as the majority (80%) of confirmed cases in HK have been mild without respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
detection of viral RNA from one or more participants' air samples | within 4 hours after starting respiratory therapy
  quantitative RTPCR from air samples

SECONDARY OUTCOMES:
the nasopharyngeal flocked swab and throat swab viral load (log10 copies/mL) | up to 2 weeks
  quantitative RTPCR from upper airway swab

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the results